CLINICAL TRIAL: NCT02251041
Title: Combined Drug Approach to Prevent Ischemia-reperfusion Injury During Transplantation of Livers (CAPITL): a First-in-men Study
Brief Title: Combined Drug Approach to Prevent Ischemia-reperfusion Injury During Transplantation of Livers (CAPITL)
Acronym: CAPITL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAPITL RCT; NCT01886443 (obsolete NCT alias)
Record Dates: First submitted 2014-09-24; First posted 2014-09-26 (Estimated); Results first posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2015-12

CONDITIONS: Reperfusion Injury
Keywords: Liver; Transplantation; Ischemia-reperfusion; Effectiveness
MeSH Terms: conditions — Reperfusion Injury | interventions — Antithrombin III; Infliximab; apotransferrin; Complement C1 Inhibitor Protein; Glutathione; Melatonin; Epoprostenol; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cases (Active Comparator): the group receives a combination of drugs
  Interventions: Drug: Antithrombin-III; Drug: Infliximab; Drug: Apotransferrin; Drug: Human recombinant erythropoietin; Drug: C1-Inhibitor; Drug: Glutathione; Drug: Alfa-tocopherol; Drug: Melatonin; Drug: Epoprostenol
- controls (Placebo Comparator): the group do not receive a combination of drugs, but a placebo (sodium chloride solution)
  Interventions: Drug: Sodium chloride solution

INTERVENTIONS:
Drug: Antithrombin-III
  Arms: cases
Drug: Infliximab
  Arms: cases
Drug: Apotransferrin
  Arms: cases
Drug: Human recombinant erythropoietin
  Arms: cases
Drug: C1-Inhibitor
  Arms: cases
Drug: Glutathione
  Arms: cases
Drug: Alfa-tocopherol
  Arms: cases
Drug: Melatonin
  Arms: cases
Drug: Epoprostenol
  Arms: cases
Drug: Sodium chloride solution
  Arms: controls

SUMMARY:
The purpose of this study is to establish the effectiveness of the combined drug approach (anti-thrombin III, infliximab, apotransferrin, human recombinant erythropoietin beta, C1-inhibitor, glutathione, alfa-tocopherol, melatonin and epoprostenol)aimed to reduce ischemia-reperfusion injury during liver transplantation in eligible recipients.

DETAILED DESCRIPTION:
This unicentric, investigator-driven, open-label randomized clinical trial with 2 parallel arms was conducted in Belgium from September 2013 through February 2018, with 1-year follow-up. Adults wait-listed for a first solitary full-size liver transplant were screened for eligibility. Exclusion criteria were acute liver failure, kidney failure, contraindication to treatment, participation in another trial, refusal, technical issues, and death while awaiting transplant. Included patients were enrolled and randomized at the time of liver offer. Data were analyzed from May 20, 2019, to May 27, 2020.

Participants were randomized to a combined drug approach with standard of care (static cold storage) or standard of care only (control group). In the combined drug approach group, following static cold preservation, donor livers were infused with epoprostenol (ex situ, portal vein); recipients were given oral α-tocopherol and melatonin prior to anesthesia and intravenous antithrombin III, infliximab, apotransferrin, recombinant erythropoietin-β, C1-inhibitor, and glutathione during the anhepatic and reperfusion phase.

The primary outcome was the posttransplant peak serum aspartate aminotransferase (AST) level within the first 72 hours. Secondary end points were the frequencies of postreperfusion syndrome, ischemia-reperfusion injury score, early allograft dysfunction, surgical complications, ischemic cholangiopathy, acute kidney injury, acute cellular rejection, and graft and patient survival.

ELIGIBILITY:
Inclusion Criteria:

1. Patients suffering from irreversible liver failure eligible for liver transplantation according to Eurotransplant guidelines.
2. Patients > 18 years of age at time of listing on Eurotransplant waiting list for liver transplantation in University Hospitals Leuven, Belgium.

Exclusion Criteria:

1. Patients who refuse to participate in the study.
2. History of hypersensitivity to one/several component(s) of the combined drug approach.
3. Conditions that prevent the use of the combined drug approach:

   * Administration of heparin at therapeutic dose pre-operatively,
   * Congestive heart failure,
   * History of seizure, poorly controlled arterial hypertension, myocardial infarction or stroke in the month preceding the liver transplantation, venous thromboembolic disease,
   * Unstable angina pectoris,
   * Sepsis, abcesses or opportunistic infections,
   * History of infliximab treatment,
   * Use of vitamin K antagonist anticoagulation.
4. Mental conditions rendering the subject incapable to understand the nature, scope, and consequences of the trial.
5. Combined organ transplantation.
6. Re-transplantation.
7. Patients that are dialysis-dependent prior to the liver transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diethard Monbaliu, MD, PhD, Principal Investigator — Abdominal transplant surgery - transplant coordination, Abdominal transplant surgery lab (microbiology & immunology Dpt)
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

REFERENCES:
- [Background] Monbaliu D, Vekemans K, Hoekstra H, Vaahtera L, Libbrecht L, Derveaux K, Parkkinen J, Liu Q, Heedfeld V, Wylin T, Deckx H, Zeegers M, Balligand E, Buurman W, van Pelt J, Porte RJ, Pirenne J. Multifactorial biological modulation of warm ischemia reperfusion injury in liver transplantation from non-heart-beating donors eliminates primary nonfunction and reduces bile salt toxicity. Ann Surg. 2009 Nov;250(5):808-17. doi: 10.1097/SLA.0b013e3181bdd787. PMID 19826248
- [Background] Vekemans K, Monbaliu D, Balligand E, Heedfeld V, Jochmans I, Pirenne J, van Pelt J. Improving the function of liver grafts exposed to warm ischemia by the Leuven drug protocol: exploring the molecular basis by microarray. Liver Transpl. 2012 Feb;18(2):206-18. doi: 10.1002/lt.22446. PMID 21987442
- [Derived] Meurisse N, Mertens M, Fieuws S, Gilbo N, Jochmans I, Pirenne J, Monbaliu D. Effect of a Combined Drug Approach on the Severity of Ischemia-Reperfusion Injury During Liver Transplant: A Randomized Clinical Trial. JAMA Netw Open. 2023 Feb 1;6(2):e230819. doi: 10.1001/jamanetworkopen.2023.0819. PMID 36853611

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 143 enrolled participants, 93 were randomized.
  Reasons for exclusion of enrolled participants was :
  * Patients deceased before transplantation (on waiting list)
  * Patients not eligible anymore for transplantation
  * Included in other clinical trials
  * Change from single liver transplantation to combined transplantation (liver-kidney)
Groups:
- Combined Drug Approach: the group receives a combination of drugs
  Antithrombin-III
  Infliximab
  Apotransferrin
  Human recombinant erythropoietin
  C1-Inhibitor
  Glutathione
  Alfa-tocopherol
  Melatonin
  Epoprostenol
- Controles: the group do not receive a combination of drugs, but a placebo (sodium chloride solution)
  Sodium chloride solution
Period: Overall Study
Arm/Group | Combined Drug Approach | Controles
Started | 53 | 40
Completed | 38 | 36
Not Completed | 15 | 4
Not completed — Did not receive intervention | 15 | 4

BASELINE CHARACTERISTICS:
Groups:
- Controls: the group do not receive a combination of drugs, but a placebo (sodium chloride solution)
  Sodium chloride solution
- Total: Total of all reporting groups
Arm/Group | Combined Drug Approach | Controls | Total
Number analyzed (Participants) | 38 | 36 | 74
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 59 [53 to 66] | 60 [51 to 68] | 60 [51 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 28 | 25 | 53
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race data were not collected from participants Population: Race data were not collected from participants
Donor age [Median (Inter-Quartile Range); unit: years] | 57 [49 to 70] | 59 [48 to 68] | 59 [48 to 69]
Donor type [Count of Participants; unit: Participants] — Donation after Circulatory Death (DCD) refers to the retrieval of organs for the purpose of transplantation from patients whose death is diagnosed and confirmed using cardio-respiratory criteria.
  Donation after Brain Death (DBD) refers to retrieval of organs for the purpose of transplantation from patients whose death is diagnosed an confirmed using neurological criteria.
  Participants
    Donation after Brain Death | 26 | 23 | 49
    Donation after Circulatory Death | 12 | 13 | 25
Warm ischemia time if Donation after Circulatory Death [Median (Inter-Quartile Range); unit: minutes] — The time between withdrawal of mechanical ventilation and abdominal aorta cannulation with initiation of cold preservation Population: Only livers from Donation after Circulatory Death donors undergo (donor) warm ischemia. So this is only measured and reported in the DCD population (see donor type)
  minutes
    number analyzed (Participants) | 12 | 13 | 25
    (all) | 17 [16 to 21] | 16 [12 to 25] | 17 [13 to 21]
Intensive Care Unit Length of stay (donor) [Median (Inter-Quartile Range); unit: days] | 3 [1 to 7] | 4 [3 to 7] | 4 [2 to 7]
Donor cause of death [Count of Participants; unit: Participants]
  Trauma | 6 | 11 | 17
  Cerebrovascular accident | 20 | 11 | 31
  Anoxia | 0 | 2 | 2
  Other | 12 | 12 | 24
Type of preservation solution [Count of Participants; unit: Participants] — Solutions used to preserve organs during storage and transport to the recipient
  Participants
    HTK (Histidine-tryptophan-ketoglutarate) | 6 | 5 | 11
    UW (University of Wisconsin) | 7 | 5 | 12
    IGL-1 (Institut Georges Lopez-1) | 25 | 25 | 50
    Other | 0 | 1 | 1
Brain death duration [Median (Inter-Quartile Range); unit: hours] — Population: The duration of brain death is only measured in Donation after Brain Death donors (see Donor type)
  hours
    number analyzed (Participants) | 26 | 23 | 49
    (all) | 13.3 [10.5 to 17.1] | 14.3 [10.0 to 20.8] | 13.5 [10.4 to 19.6]
Donor hepatectomy duration [Median (Inter-Quartile Range); unit: minutes] | 34.5 [25.0 to 46.0] | 32.5 [26.0 to 42.5] | 34 [25.5 to 43.8]
Cold ischemia time [Median (Inter-Quartile Range); unit: hours] — Time from start of cold flush until the organ leaves the ice and is placed in the body of the recipient
  hours | 5.8 [4.8 to 8.1] | 5.8 [5.1 to 8.1] | 5.8 [5.0 to 8.0]
Model for End-Stage Liver Disease score (MELD) [Median (Inter-Quartile Range); unit: score on a scale] — Model for End-Stage Liver Disease score is a score based on bilirubin, creatinine and INR to calculate the severity of liver disease. The score ranges from 6 tot 40 and the higher the number the more likely you are to receive a liver from a deceased donor when an organ becomes available.
  score on a scale | 13.2 [8.7 to 19.1] | 13.8 [10.8 to 19.4] | 13.6 [10.2 to 19.2]
Indication for liver transplant [Number; unit: participants] — Patients can have multiple indications for transplantation
  participants
    Metabolic disease | 4 | 3 | 7
    HCC | 18 | 12 | 30
    Chronic liver disease | 25 | 18 | 43
    Ethyl | 23 | 18 | 41
    HBV | 2 | 0 | 2
    HCV | 2 | 0 | 2
    Cholestatic disease | 4 | 4 | 8
    Nonalcoholic Steatohepatitis | 2 | 10 | 12
    Cryptogenic | 1 | 0 | 1
Implantation duration [Median (Inter-Quartile Range); unit: Minutes] — Implantation duration is the time between the organ leaving the ice box and the restoration of the blood supply in the recipient.
  Minutes | 39.5 [35.0 to 48.0] | 38.5 [34.5 to 45.0] | 39.0 [35.0 to 45.0]

OUTCOME MEASURES:

1. Primary Outcome: Peak Aspartate Aminotransferase Within First 72h Post Transplant
Description: peak AST is defined as the highest value of serum AST within 72 hours following liver transplantation
Time Frame: within 72 hours following liver transplantation
Measure: Geometric Mean (95% Confidence Interval); unit: U/L
Arm/Group | Combined Drug Approach | Controles
Number analyzed (Participants) | 36 | 36
U/L | 1262.9 [946.3 to 1685.4] | 1451.2 [1087.4 to 1936.7]

2. Secondary Outcome: Graft Loss
Description: graft loss at 3 and 12 months after liver transplantation
Time Frame: 3 and 12 months after liver transplantation
Population: Death-censored graft survival
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Drug Approach | Controles
Number analyzed (Participants) | 36 | 36
Participants
  3-months | 2 | 0
  12-months | 3 | 0

3. Secondary Outcome: Recipient Death
Description: recipient death at 3 and 12 months after liver transplantation
Time Frame: 3 and 12 months after liver transplantation
Measure: Count of Participants; unit: Participants
Groups:
- Cases: the group receives a combination of drugs
  Antithrombin-III
  Infliximab
  Apotransferrin
  Human recombinant erythropoietin
  C1-Inhibitor
  Glutathione
  Alfa-tocopherol
  Melatonin
  Epoprostenol
Arm/Group | Cases | Controles
Number analyzed (Participants) | 36 | 36
Participants
  3 months | 3 | 1
  12 months | 4 | 3

4. Secondary Outcome: Early Graft Dysfunction
Description: early graft dysfunction as defined by Olthoff
Time Frame: within first 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Cases | Controles
Number analyzed (Participants) | 36 | 36
Participants | 13 | 17

5. Secondary Outcome: Number of Participants Developing Biliary Strictures
Description: Biliary strictures are the narrowing of the intrahepatic or extrahepatic biliary ductal system. Here we report the number of participants developing biliary strictures within 12 months post transplantation by MRCP (magnetic resonance cholangiopancreatography)
Time Frame: within 12 months post transplantation
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Drug Approach | Controles
Number analyzed (Participants) | 36 | 36
Participants | 13 | 10

6. Secondary Outcome: Ischemia Reperfusion Injury Score
Description: Ischemia Reperfusion Injury score 1h post reperfusion by using the Suzuki score and Monbaliu et al. The score ranges from 0 (no injury) to 4 (severe injury).
Time Frame: One hour post reperfusion
Measure: Median (Inter-Quartile Range); unit: score
Arm/Group | Combined Drug Approach | Controles
Number analyzed (Participants) | 25 | 23
score | 2 [2 to 4] | 2 [1 to 4]

7. Secondary Outcome: Graft Rejection
Description: a liver biopsy will be taken after transplantation and in case of clinical suspicion of acute rejection
Time Frame: till 1 year after transplantation
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Drug Approach | Controles
Number analyzed (Participants) | 36 | 36
Participants | 9 | 8

8. Secondary Outcome: Patients With at Least 1 Severe Surgical Complications
Description: The ranking of surgical complications will be done by using Clavien-Dindo classification
  Grade I Any deviation from the normal post-operative course not requiring surgical, endoscopic or radiological intervention. This includes the need for certain drugs (e.g. antiemetics, antipyretics, analgesics, diuretics and electrolytes), treatment with physiotherapy and wound infections that are opened at the bedside Grade II Complications requiring drug treatments other than those allowed for Grade I complications; this includes blood transfusion and total parenteral nutrition (TPN) Grade III Complications requiring surgical, endoscopic or radiological intervention Grade IV Life-threatening complications; this includes CNS complications (e.g. brain haemorrhage, ischaemic stroke, subarachnoid haemorrhage) which require intensive care, but excludes transient ischaemic attacks (TIAs) Grade V Death of the patient
  A severe surgical complication is defined as Grade III or higher.
Time Frame: within 1 year after liver transplantation
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Drug Approach | Controles
Number analyzed (Participants) | 36 | 36
Participants | 10 | 8

9. Secondary Outcome: Non-anastomotic Biliary Stricture
Description: Non-anastomotic biliary stricture at 1 year
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Drug Approach | Controles
Number analyzed (Participants) | 36 | 36
Participants | 4 | 2

10. Secondary Outcome: Acute Kidney Injury Score
Description: An acute kidney injury score of 1 indicates risk; 2, injury; and 3, failure. According to RIFLE (Risk, Injury, Failure, Loss of kidney function, and End-stage kidney disease) Minimum score is 0 meaning there is no injury, maximum score is 3 meaning failure of the organ.
Time Frame: 48h
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Drug Approach | Controles
Number analyzed (Participants) | 34 | 35
Participants
  RIFLE 0 | 27 | 31
  RIFLE 1 | 4 | 1
  RIFLE 2 | 2 | 3
  RIFLE 3 | 1 | 0

11. Secondary Outcome: Post-Reperfusion Syndrome
Description: Post-reperfusion syndrome defined as a 30% decrease of mean systemic blood pressure for more than 1 minute during the first 5 minutes following graft reperfusion
Time Frame: first 5 minutes following graft reperfusion
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Drug Approach | Controles
Number analyzed (Participants) | 29 | 29
Participants | 7 | 6

12. Other Pre Specified Outcome: Intensive Care Unit Length of Stay (Recipient)
Description: Intensive Care Unit stay immediately after liver transplantation (not after rehospitalization)
Time Frame: During hospital stay for liver transplantation
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Combined Drug Approach | Controles
Number analyzed (Participants) | 38 | 36
Days | 3 [1.5 to 6.5] | 4 [2.5 to 7.0]

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the time frame of 1 year starting immediately after transplantation
Arm/Group | Combined Drug Approach | Controles
All-Cause Mortality (participants affected / at risk) | 4/36 | 3/36
Serious Adverse Events (participants affected / at risk) | 6/36 | 4/36
Other Adverse Events (participants affected / at risk) | 33/36 | 31/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Combined Drug Approach (N=36) | Controles (N=36)
General surgical complications (Surgical and medical procedures) | 2 | 2
Respiratory insufficiency (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Kidney dysfunction (Renal and urinary disorders) | 1 | 0
Bacterial infection (Infections and infestations) | 1 | 0
Arrythmia (Cardiac disorders) | 1 | 0
Portal vein thrombosis (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Combined Drug Approach (N=36) | Controles (N=36)
Post-operative delirium (General disorders) | 9 | 11
Acute kidney injury (Renal and urinary disorders) | 12 | 9
Respiratory failure post-op (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Urinary tract infections (Renal and urinary disorders) | 2 | 5
De novo diabetes mellitus (Endocrine disorders) | 3 | 2
Viral infections (Infections and infestations) | 6 | 1
Bacterial infections (Infections and infestations) | 16 | 10
Fungal infection (Infections and infestations) | 3 | 3
Thrombo-embolitic complications (Blood and lymphatic system disorders) | 0 | 2
Cardiovascular events (Cardiac disorders) | 2 | 6
Cerebrovascular events (General disorders) | 0 | 1
Organ specific complications (Hepatobiliary disorders) | 5 | 6
Surgical complications - arterial (Injury, poisoning and procedural complications) | 2 | 2
Surgical complications portal (Injury, poisoning and procedural complications) | 2 | 3
Surgical complications - general (Injury, poisoning and procedural complications) | 22 | 18
Biliary problems (Hepatobiliary disorders) | 6 | 5
Rejections (Immune system disorders) | 6 | 6

LIMITATIONS AND CAVEATS:
* Single center RCT
* Individual effects of each component of CDA in decreasing IRI were not assessed separately.
* Despite the fact that CDA components were administrated according to a specific timing in relation to their pharmacokinetics with the aim to reach a peak concentration during reperfusion, blood levels of each component were not determined.
* Although the study was powered to detect differences in peak AST, the small sample size did not allow a claim on the absence of an effect.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-08): https://cdn.clinicaltrials.gov/large-docs/41/NCT02251041/Prot_SAP_000.pdf